CLINICAL TRIAL: NCT03918421
Title: Immunoglobulin M (IgM)-Anti-myelin-associated-glycoprotein(MAG) Peripheral Neuropathy Study: From Proper Assessment to Trial Needs - IMAGiNe Study-Lyon/Bicêtre
Brief Title: Immunoglobulin M (IgM)-Anti-myelin-associated-glycoprotein(MAG) Peripheral Neuropathy Study
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0217; 2019-A00884-53 (Other: ID-RCB)
Record Dates: First submitted 2019-04-15; First posted 2019-04-17 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Immunoglobin M Anti-myelin-associated-glycoprotein Peripheral Neuropathy
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Immunogloblin M-anti myelin-associated-glycoprotein neuropathy: Patient group (25 subjects) presenting with an Immunogloblin M-anti myelin-associated-glycoprotein peripheral neuropathy
  Interventions: Other: Clinical examination and patients' questionnaires regarding activity and participation (preliminary Immunogloblin M (IgM)-Rasch-built overall Disability Scale (RODS), and finalized IgM-RODS)

INTERVENTIONS:
Other: Clinical examination and patients' questionnaires regarding activity and participation (preliminary Immunogloblin M (IgM)-Rasch-built overall Disability Scale (RODS), and finalized IgM-RODS) — Rasch-built overall Disability Scale (RODS) is a disease-specific, patient-based, linearly weighted scale that captures activity and social participation limitations to detect activity limitations in patients with Immunogloblin M (IgM) anti-myelin-associated-glycoprotein peripheral neuropathy. For this study, the preliminary RODS is a 146 item patient-reported outcome instrument that assesses activity and social participation limitation. Rasch Measurement Methods examine the extent observed data (patients' actual responses to scale items) accord with predictions of those responses from a mathematical model.

SUMMARY:
There is no international consensus regarding how to assess and treat patients with immunoglobulin M (IgM)-anti-myelin-associated-glycoprotein (MAG) monoclonal gammopathy associated peripheral neuropathy. The purpose of the IMAGiNe study-Lyon/Bicêtre is to prospectively collect standardized clinical data of 25 patients with IgM-anti-MAG monoclonal gammopathy associated peripheral neuropathy in order to participate in the international IMAGiNe Study.

The main objective is to describe in detail the various clinical subtypes, clinical course, treatment responses, antibody titers of IgM-anti-MAG monoclonal gammopathy associated peripheral neuropathy using a variety of outcome measures. The obtained observational data will allow the construction of an IgM monoclonal gammopathy associated peripheral neuropathy-specific Rasch-built overall Disability Scale (RODS) that should fulfill all modern clinimetric requirements, including cross-cultural validity. The coordinating centers for the IgM-RODS construction will be the Maastricht University Medical Center and University Medical Center Utrecht, both in the Netherlands.

ELIGIBILITY:
Inclusion Criteria:

* fulfilling the international criteria for the diagnosis Immunogloblin M (IgM) monoclonal gammopathy, with anti-myelin-associated-glycoprotein (MAG) antibodies, and peripheral neuropathy.
* age of 18 years or older followed in neuromuscular department of Lyon;
* informed consent given by the participant

Exclusion Criteria:

* concomitant diseases possibly interfering with peripheral nerve and function, as well as physical functioning, such as diabetes, renal insufficiency, (prior) treatment with chemotherapy for diseases other than their Immunogloblin M (IgM) monoclonal gammopathy associated peripheral neuropathy, history of hereditary neuropathy, vitamin deficiency, connective tissue disorder, hepatitis B and C and human immunodeficiency virus (HIV) infection, alcohol abuse (more than 5 International Units(IU)/day);
* an active malignancy with poor prognosis, undergoing treatment aside from monoclonal gammopathy associated peripheral neuropathy;
* pregnant;
* the use of any medication that may cause peripheral nerve function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at least 18 years old fulfilling the international criteria for Immunogloblin M (IgM)-anti-myelin-associated-glycoprotein (MAG) monoclonal gammopathy and peripheral neuropathy
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2020-06-23 (Actual); Primary Completion 2030-06-23 (Estimated); Study Completion 2030-06-23 (Estimated)

PRIMARY OUTCOMES:
Change in patient activity and participation according to patient questionnaires | 0, 6, 12, 24 and 36 months
  Preliminary Immunogloblin M (IgM)-Rasch-built Overall Disability Scale (RODS), and after its construction the finalized IgM-RODS. Rasch-built overall Disability Scale (RODS) is a disease-specific, patient-based, linearly weighted scale that captures activity and social participation limitations to detect activity limitations in patients with Immunogloblin M (IgM) anti-myelin-associated-glycoprotein peripheral neuropathy. For this study, the preliminary RODS is a 146 item patient-reported outcome instrument that assesses activity and social participation limitation. Rasch Measurement Methods examine the extent observed data (patients' actual responses to scale items) accord with predictions of those responses from a mathematical model.

CONTACTS AND LOCATIONS:
Overall Officials: Juliette SVAHN, MD, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Hospices Civils de Lyon Service Neurologie C, Pathologies Neuromusculaires, Unité 302, Bron
  - Centre de référence NNERf, Le Kremlin-Bicêtre